CLINICAL TRIAL: NCT02172079
Title: Effects of Mobilization-with-Movement on Pain and Range of Motion in Unilateral Shoulder Impingement Syndrome: A Randomized Controlled Trial
Brief Title: Mobilization With Movement for Shoulder Impingement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: César Fernández-de-las-Peñas (Other)
Collaborators: University of Salamanca (Other)
Responsible Party: Sponsor-Investigator, César Fernández-de-las-Peñas, Proffesor, Universidad Rey Juan Carlos
Organization: Universidad Rey Juan Carlos (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: USAL201000048540
Record Dates: First submitted 2014-06-22; First posted 2014-06-24 (Estimated); Last update posted 2014-06-24 (Estimated); Status verified 2014-06

CONDITIONS: Shoulder Impingement Syndrome
Keywords: shoulder impingement, manual therapy, pain, motion.
MeSH Terms: conditions — Shoulder Impingement Syndrome; Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Real mobilization-with-movement (MWM) (Experimental): For the MWM group, an accessory posterior-lateral gliding movement in the humeral head combined with a movement of active shoulder flexion will be applied. One hand will be placed over the scapula posteriorly while the thenar eminence of the other hand will be placed over the anterior aspect of the head of the humerus
  Interventions: Other: Real mobilization-with-movement (MWM)
- Sham mobilization-with-movement (MWM) (Sham Comparator): The sham condition will replicate the treatment condition except for the hand positioning. The therapist locates one hand over the belly of the pectoralis major muscle and the other over scapula without applying any pressure. The patient will be asked to move the arm in a similar manner as in the MWM group
  Interventions: Other: Sham mobilization-with-movement (MWM)

INTERVENTIONS:
Other: Real mobilization-with-movement (MWM)
  Arms: Real mobilization-with-movement (MWM)
Other: Sham mobilization-with-movement (MWM)
  Arms: Sham mobilization-with-movement (MWM)

SUMMARY:
Controversy exists regarding the effectiveness of manual therapy techniques for the management of impingement syndrome. However, no adequately powered clinical trials have examined the effects of mobilization-with-movement. The purpose of the current study was to perform a randomized controlled trial comparing the effects of real MWM to a group receiving a sham intervention on shoulder pain at different moments and active shoulder range of motion in an adequately powered sample of patients with shoulder impingement syndrome.

ELIGIBILITY:
Inclusion Criteria:

* history of shoulder pain of > 3months duration
* pain localized at the proximal anterolateral shoulder region
* medical diagnosis of shoulder impingement syndrome
* at least 2 positive impingement tests including Neer, Hawking, or Jobe test

Exclusion Criteria:

* diagnosis of fibromyalgia
* pregnancy
* a history of traumatic onset of shoulder pain
* other histories of shoulder injury
* ligamentous laxity based on a positive Sulcus test and apprehension test
* numbness or tingling in the upper extremity
* previous shoulder or cervical spine surgery
* corticosteroid injection on the shoulder within 1 year of the study
* physical therapy 6 months prior to the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2013-01; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Changes in the intensity of shoulder pain before and after the treatment | Baseline and one week after intervention
  Participants were asked to rate the intensity of their pain using an 11-point numerical pain rating scale (NPRS; 0: no pain; 10: maximum pain) for 3 scores of perceived pain: 1, the intensity of shoulder pain experienced in the last 24h; 2, the intensity of shoulder pain at night; 3, the intensity of shoulder pain during shoulder flexion.

SECONDARY OUTCOMES:
Changes in shoulder range of motion before and after the treatment | Baseline and one week after the intervention
  A universal goniometer was used to assess the participant's shoulder range of motion in the following motions:
  * Pain-free and maximum (painful) range of motion in shoulder flexion
  * Pain-free range of motion in shoulder extension
  * Pain-free range of motion in shoulder abduction
  * Pain-free range of motion in shoulder external rotation
  * Pain-free range of motion in shoulder medial (internal) rotation

CONTACTS AND LOCATIONS:
Overall Officials: Francisco Alburquerque Sendín, PT, PhD, Principal Investigator — University of Salamanca; César Fernández de las Peñas, PT, PhD, Study Chair — Universidad Rey Juan Carlos
Locations (1):
- Francisco Alburquerque Sendín, Salamanca, Salamanca, Spain